CLINICAL TRIAL: NCT03174756
Title: EVALUATION OF THE HYPOCHLOROUS ACID SUBSTANTIVITY AS ANTI-PLAQUE AGENT. A RANDOMIZED CONTROLLED TRIAL
Brief Title: HYPOCHLOROUS ACID SUBSTANTIVITY AS ANTIPLAQUE AGENT (HOCl-SAP)
Acronym: HOCl-SAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad El Bosque, Bogotá (Other)
Responsible Party: Principal Investigator, Gloria Inés Lafaurie, Magister Clinical Epidemiology, Universidad El Bosque, Bogotá
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ubosque
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Hypochlorous Acid; Mouthwashes
Keywords: Hypochlorous Acid; Chlorhexidine; Antiplaque agents; Substantivity
MeSH Terms: interventions — Hypochlorous Acid; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: A double-blind randomized controlled trial with 75 participants was conducted. Participants were assigned using block randomization in five groups: HOCl 0.025% and 0.05%, CHX 0.12% and 0.2% and sterile water as placebo. Participants were instructed to use each rinse solution for 30 seconds after dental prophylaxis. Samples of saliva were taken at baseline and after 30 seconds, 1, 3.5 and 7 hours to assess substantivity establishing the bacterial viability by the fluorescence method.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The treatment codes of the study were not accessible to the investigators and to the examiner until the data were analyzed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- HOCl 0.025% (Experimental): 15 ml of Hypochlorous acid mouthwash at 0.025%
  Interventions: Drug: Hypochlorous Acid
- HOCl 0.05% (Experimental): 15 ml of Hypochlorous acid mouthwash at 0.05%
  Interventions: Drug: Hypochlorous Acid
- CHX 0.2% (Active Comparator): 15 ml of chlorhexidine mouthwash at 0.2%
  Interventions: Drug: Chlorhexidine
- CHX 0.025% (Active Comparator): 15 ml of chlorhexidine at mouthwash0.025%
  Interventions: Drug: Chlorhexidine
- Placebo (Placebo Comparator): 15 ml of Sterile water
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hypochlorous Acid — Mouthwashes of antiplaque agents
  Other Names: HClO; Hypochlorous Acids
  Arms: HOCl 0.025%; HOCl 0.05%
Drug: Chlorhexidine — A disinfectant and topical anti-infective agent used also as mouthwash to prevent oral plaque.
  Other Names: CHX
  Arms: CHX 0.025%; CHX 0.2%
Other: Placebo — Sterile water as placebo
  Other Names: Placebos
  Arms: Placebo

SUMMARY:
Hypochlorous acid (HOCl) in a non-antibiotic antimicrobial agent used in clinical medicine. Nevertheless, its antiplaque oral effect has not been evaluated. Chlorhexidine (CHX) is the gold standard as an antiplaque agent for its high substantivity in plaque and saliva. There are no published studies evaluating the substantivity of hypochlorous acid compared to CHX. Objective: To evaluate the efficacy of mouthwashes of HOCl in substantivity evaluated by reduction of bacterial viability in saliva during 7 hours compared to CHX rinses and a placebo.

DETAILED DESCRIPTION:
Materials and Methods: A randomized, double-blind clinical trial with 75 participants was conducted. Participants were randomly assigned using block randomization in five groups: HOCl 0.025% and 0.05%, CHX 0.12 and 0.2% and sterile water as placebo. Participants were instructed to use each rinse with 10 ml of each solution for 30 seconds after dental prophylaxis. Samples of saliva were taken at baseline and after 30 seconds, 1, 3.5 and 7 hours to assess substantivity establishing the bacterial viability by the fluorescence method with the SYTO 9/propidium iodide dual staining. All participants were assessed with the Turesky visible plaque index at baseline and at 7 hours and adverse events were assessed. For the comparisons of the viability of the different rinses between times, the statistical test of generalized linear mixed model [GT1] adjusted to treatment, time and treatment-time interaction was used.

ELIGIBILITY:
Inclusion Criteria:

* Dentate young men with minimum 22 teeth were considered eligible for the study. Participants should have good dental and gingival status (DMFT index ≤ 3, median of Lobene gingival index ≤ 1) and detectable levels of dental plaque at 7 hours of brushing during the selection process.

Exclusion Criteria:

* Exclusion criteria included smoking, orthodontic, orthopedic or rehabilitation treatment, cavitated carious lesions and consumption of systemic antimicrobials or anti-inflammatory drugs in the last 6 months.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Substantivity | Baseline, 30 Seconds, 1, 3, 5 and 7 hours
  Viability reduction (VR) was calculated for each saliva sample by the difference in the percentage of viable bacteria between two times.

SECONDARY OUTCOMES:
Plaque Index | Baseline and 7 hours
  Visible plaque was evaluated by Turesky Index 1970

OTHER OUTCOMES:
Adverse effect | 24 hours
  A survey was applied to each of the patients in order to record if any adverse effects occurred after the use of each of the interventions as burning and pain in the oral mucosa and was investigated by the taste of substances and sensation of dryness. An examiner evaluated the buccal, labial, lingual, pharyngeal and teeth tissues to establish changes and alterations visible to the clinical examination and the presence of candidiasis.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Ines Lafaurie, MS, Principal Investigator — El Bosque University
Locations (1):
- Gloria Ines Lafaurie, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No
No requerid

REFERENCES:
- [Result] Lafaurie GI, Calderón JL, Zaror C, Millán LV, Castillo DM. Hypochlorous Acid: A New Alternative as Antimicrobial Agent and For Cell Proliferation for Use in Dentistry. International journal of odontostomatology. 9: 475-481. 2015
- [Result] Castillo DM, Castillo Y, Delgadillo NA, Neuta Y, Jola J, Calderon JL, Lafaurie GI. Viability and Effects on Bacterial Proteins by Oral Rinses with Hypochlorous Acid as Active Ingredient. Braz Dent J. 2015 Oct;26(5):519-24. doi: 10.1590/0103-6440201300388. PMID 26647939
- [Result] Chen CJ, Chen CC, Ding SJ. Effectiveness of Hypochlorous Acid to Reduce the Biofilms on Titanium Alloy Surfaces in Vitro. Int J Mol Sci. 2016 Jul 19;17(7):1161. doi: 10.3390/ijms17071161. PMID 27447617
- [Result] Moran J, Addy M, Wade W, Milson S, McAndrew R, Newcombe RG. The effect of oxidising mouthrinses compared with chlorhexidine on salivary bacterial counts and plaque regrowth. J Clin Periodontol. 1995 Oct;22(10):750-5. doi: 10.1111/j.1600-051x.1995.tb00257.x. PMID 8682921
- [Result] Wang L, Bassiri M, Najafi R, Najafi K, Yang J, Khosrovi B, Hwong W, Barati E, Belisle B, Celeri C, Robson MC. Hypochlorous acid as a potential wound care agent: part I. Stabilized hypochlorous acid: a component of the inorganic armamentarium of innate immunity. J Burns Wounds. 2007 Apr 11;6:e5. PMID 17492050